CLINICAL TRIAL: NCT06412874
Title: Assessment of Supportive Care and Educational Needs to Guide Quality Care Improvements for Patients With Locally Advanced and Metastatic Bladder Cancer
Acronym: ACCESS
Status: Active, not recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Nihal E Mohamed, Nihal Mohamed, Associate Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: STUDY-23-00592
Record Dates: First submitted 2023-10-09; First posted 2024-05-14 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-08

CONDITIONS: Screening Tool; Focus Group
MeSH Terms: interventions — Potentially Inappropriate Medication List

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Screening tool group
  Interventions: Other: Screening tool
- Focus group

INTERVENTIONS:
Other: Screening tool — Participants will complete a screening tool survey
  Groups: Screening tool group

SUMMARY:
The overall goal of this study is to facilitate care improvements for bladder cancer patients with locally advanced or metastatic disease by designing and evaluating a patient need assessment screening tool to be used, in the future, as standard screening measure. Adult individuals diagnosed with Stage 4 incurable locally advanced or metastatic bladder cancer will be included in this study and asked to participate in a focus group, complete a screening tool, or complete a survey. All data collected will be linked to a study ID number and HIPAA identifiers will not be linked to study data. Identifying information (ie: name, mrn, email, phone number) will be utilized for study recruitment and identifying eligible patients. Any disclosure of the human subjects' responses outside the research would not reasonably place the subjects at risk of criminal or civil liability or be damaging to the subjects' financial standing, employability, educational advancement, or reputation.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible to participate if they are diagnosed with Stage 4 incurable locally advanced or metastatic bladder cancer
* between 18 years and older (18-89 years)
* have initiated any systemic treatment for advanced urothelial carcinoma
* speak English speaking and are able to consent.

Exclusion Criteria:

* Have a diagnosis of another advanced cancer that has required systemic therapy
* Or have any condition that, in the opinion of the investigator, would compromise the well- being of the subject or the study or prevent the subject from meeting or performing study requirements.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bladder cancer survivors
Sampling Method: Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
The Bladder Cancer Need Assessment Survey (BCNAS) | 2023-2025
  The Bladder Cancer Need Assessment Survey (BCNAS) includes 8 subscales: psychological, informational, care and support, logistic, sexuality, physical and daily living, communication with providers; and communication with social partners/family
  All subscales scored 0-100. Full scale scored from 0- 100. Higher score mean higher levels of unmeet needs.
  This is a measure of unmet needs.

CONTACTS AND LOCATIONS:
Overall Officials: Nihal Mohamed, PhD, Principal Investigator — Icahn School of Medicine
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No